CLINICAL TRIAL: NCT01213875
Title: A Multifaceted Nurse-based Strategy Reduces HEart FaiLure Morbidity in PatiENts Admitted for Acute Decompensated Heart Failure in Brazil
Acronym: HELEN II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Eneida Rejane Rabelo da Silva, Professor; PhD., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS and HCPA 09112
Record Dates: First submitted 2009-11-09; First posted 2010-10-04 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure
Keywords: heart failure; nursing; home based intervention; cost; efficacy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Intervention and control (Experimental): I: Experimental Routine monitoring by health team in the reference institution, four home visits and four telephone contacts with trained nurses.
  II: Control Routine monitoring by health team in the reference institution.
  Interventions: Behavioral: Home based education
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Home based education — There will provided education about what is heart failure, its causes, how to recognize signs and symptoms, monitoring of weight and blood pressure, the importance of compliance to treatment. Patients will be instructed about the medications; a guide to rest and exercise, sexual activity, vaccines, travel and diet will be provided. The involvement of the family will be encouraged; the contact with the team should be done when: patient observes an increase of 1 or 2 kg of weight in 2-3 days, worsening of dyspnea on effort, edema in legs / abdomen, worsening of cough, persistent vomiting, syncope,sputum with blood, fever, persistent tachycardia. In phone calls made between home visits, the compliance to treatment will be evaluated and reinforced.
  Other Names: Education on Heart Failure; Home Intervention
  Arms: Experimental: Intervention and control

SUMMARY:
The home based intervention is a multidisciplinary approach that has shown benefit in the follow-up of patients with Heart Failure (HF). It is considered one of the most effective approaches and humanized by education and care for the patient in his environment of routine. In this study the monitoring of HF patients in the home after hospital discharge will include the reinforcement, monitoring and reassessment of previously provided guidance on the disease and self-care, compliance to prescribed medications and especially the early recognition of signs and symptoms of decompensation by patients and their caregivers.

DETAILED DESCRIPTION:
The epidemiological picture of cardiovascular disease in which the IC sets itself as the leading cause of readmissions in the National Health System and that has not changed over the years, undertake the management of the limited resources of the public health system. Moreover, the IC contributes to significant loss of quality of life of patients, many in socially productive ages resulting in absenteeism and early retirement. This study aims to evaluate the impact of home monitoring, intercalated with telephone contact by the nursing staff at the HF patients, after hospital discharge in relation to the rate of hospital readmissions, compliance and cost-effectiveness this intervention, compared to conventional monitoring of patients within 6 months without this intervention, as well as building a structure that allows the use computerized forms of assessment in nursing in cardiology by mobile technology, assess the knowledge of the disease and the skills to self-care; assess compliance, assess the quality of life, linking the sociodemographic characteristics and clinical with adherence to treatment and rates of readmission in both groups, and check the cost of home monitoring. For this purpose, a randomized clinical trial was designed in two centers, blinded to outcomes and costs of readmission.

Summary of the study:

The home based intervention is a multidisciplinary approach that has shown benefit in the follow-up of patients with Heart Failure (HF). It is considered one of the most effective approaches and humanized by education and care for the patient in his environment of routine. In this study the monitoring of HF patients in the home after hospital discharge will include the reinforcement, monitoring and reassessment of previously provided guidance on the disease and self-care, compliance to prescribed medications and especially the early recognition of signs and symptoms of decompensation by patients and their caregivers.

Detailed description: The epidemiological picture of cardiovascular disease in which the IC sets itself as the leading cause of readmissions in the National Health System and that has not changed over the years, undertake the management of the limited resources of the public health system. Moreover, the IC contributes to significant loss of quality of life of patients, many in socially productive ages resulting in absenteeism and early retirement. This study aims to evaluate the impact of home monitoring, intercalated with telephone contact by the nursing staff at the HF patients, after hospital discharge in relation to the rate of hospital readmissions, compliance and cost-effectiveness this intervention, compared to conventional monitoring of patients within 6 months without this intervention, as well as building a structure that allows the use computerized forms of assessment in nursing in cardiology by mobile technology, assess the knowledge of the disease and the skills to self-care; assess compliance, assess the quality of life, linking the sociodemographic characteristics and clinical with adherence to treatment and rates of readmission in both groups, and check the cost of home monitoring. For this purpose, a randomized clinical trial was designed in two centers, blinded to outcomes and costs of readmission.

Intervention: There will provided education about what is heart failure, its causes, how to recognize signs and symptoms, monitoring of weight and blood pressure, the importance of compliance to treatment. Patients will be instructed about the medications they are using. A guide to rest and exercise, sexual activity, vaccines, travel and diet (water and salt restriction) will be provided. The involvement of the family will be encouraged and reinforced at every home visit. The contact with the team should be done when: patient observes an increase of 1 or 2 kg of weight in 2-3 days, worsening of dyspnea on effort, edema in legs / abdomen, worsening of cough, persistent vomiting, syncope, sputum with blood, fever, persistent tachycardia, motor deficit / paralysis and / or unexplained chest pain. In phone calls made between home visits, the compliance to treatment will be evaluated and reinforced.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 years or above, with a diagnosis of heart failure with systolic dysfunction (ejection fraction ≤ 45%), hospitalized for decompensation of HF
* Who agree to participate in the study by signing the Informed Consent.

Exclusion Criteria:

* Patients with communication disabilities and people with degenerative neurological diseases.
* Are also excluded patients who presented acute coronary syndrome (ACS) in the last 6 months before randomization
* Patients with renal, hepatic, pulmonary or systemic disease that may confuse the interpretation of the findings or result in limited life expectancy
* Surgical plan or therapeutic that might influence the follow-up
* Pregnancy, diagnosis of acute heart failure secondary to:

  * sepsis
  * myocarditis
  * myocardial infarction
  * acute peripartum and other cause
* Have no interest in receiving home visits
* Living at a distance greater than 10 km from the hospital of origin
* Not be able to contact by telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome was a composite end-point of a first visit to the emergency department (lasting less than 24 hours), or a first hospital readmission (> 24h) or all-cause death, assessed during the first 6 months of follow-up. | Up to 36 months.
  This primary outcomes will be measured at each visit, which will have different intervals, according to the research protocol, with a final evaluation after the last home visit.
  Home visits (HV): 7 days after discharge, 15 days after 1st phone call (PC), 30 days after 2nd PC, 30 days after 3rd PC.
  Phone calls (PC): 7-10 days after 1st HV, 30 days after 2nd HV, 30 days after 3rd HV, 15 days after 4th HV.
  All patients come to Hospital evaluation after the 4th phone call.

SECONDARY OUTCOMES:
Cost-effectiveness of visits to the emergency department and length of hospitalization. | up to 36 months
  Costs for intervention group include time of nurses home visit and telephone contacts. The effectiveness will be assessed in life earned years.
  Home visits (HV): 7 days after discharge, 15 days after 1st phone call (PC), 30 days after 2nd PC, 30 days after 3rd PC.
  Phone calls (PC): 7-10 days after 1st HV, 30 days after 2nd HV, 30 days after 3rd HV, 15 days after 4th HV.
  All patients come to Hospital evaluation after the 4th phone call.
The secondary outcomes were each individual end-points | 36 months
  All end-points were prospectively evaluated by a researcher that was blinded to group assignment, based on the final 6-months visit and the revision of available electronic records. Whenever it was not available, validation was also based on clinical discharge notes (from emergency departments or hospitals distinct from the institution of origin).

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, RN, ScD, Principal Investigator — HCPA and UFRGS
Locations (1):
- Universidade Federal do Rio Grande do Sul - Post Graduated Program, Porto Alegre, Rio Grande do Sul, Brazil